CLINICAL TRIAL: NCT05349565
Title: Effects of Muscle Energy Technique Along Conventional Physical Therapy After Mesenchymal Stem Cell Transplantation in Knee Osteoarthritis Patients
Brief Title: Effects of Muscle Energy Technique in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01255 Fanila Ashraf
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Mesenchymal stem cells (MSCs),; muscle energy technique (MET),; rehabilitation protocol
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONVENTIONAL PHYSICAL THERAPY (Active Comparator): TENS , Open chain knee flexion and extension, Calf stretch , Quad set
  Interventions: Other: CONVENTIONAL PHYSICAL THERAPY
- MUSCLE ENERGY TECHNIQUE (Experimental): MET ( isometric contraction with 6-10 sec )
  Interventions: Other: MUSCLE ENERGY TECHNIQUE

INTERVENTIONS:
Other: CONVENTIONAL PHYSICAL THERAPY — High frequency TENS for 10 mins, 3 days/week Ankle pumps for blood circulation 10 repetitions x1 set, 3 days/week. Heel slides10 repetitions x1 set, 3 days/week. Open chain knee flexion and extension 10 repetitions x1 set, 3 days/week. SLR (straight leg raise) 10 repetitions x1 set, 3 days/week. Calf stretch 10 repetitions x1 set, 3 days/week. Quad set 10 repetitions x1 set, 3 days/week.
  Total 6 sessions each consisting of 30-45 minutes
  Arms: CONVENTIONAL PHYSICAL THERAPY
Other: MUSCLE ENERGY TECHNIQUE — Experimental group treated by applying Muscle energy technique along conventional physical therapy.
  For MET patient is positioned at maximal comfort and lengthening while engaging the barrier and then patient is asked to perform isometric contraction with 6-10 sec hold and then release and lengthen the muscle 4-5 repetition x 1 set, 3days/week Total 6 sessions each consisting of 30-45 minutes
  Arms: MUSCLE ENERGY TECHNIQUE

SUMMARY:
To determine the effectiveness of muscle energy technique along conventional physical therapy after mesenchymal stem cell transplantation in knee Osteoarthritis patients regarding Pain, range of motion, functional disability and quality of life.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) replacement is a regenerative therapeutic procedures for the early treatment of cartilaginous defects in knee osteoarthritis. MSCs may improve symptoms and function in osteoarthritic joints but also decrease inflammation and induce cartilage healing by differentiating into chondrocytes, osteoblasts and indicating appropriate extracellular matrix proteins (i.e. collagen I and II) through the secretion of cytokines, chemokines, and growth factors from MSCs.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age > 40 years
* Knee osteoarthritis patients undergone mesenchymal stem cell transplantation.

Exclusion Criteria:

* History of recent or past septic arthritis
* Patients with neurological deficit
* Uncontrolled diabetes
* Malignancy
* Vascular insufficiency

Ages: 41 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | NPRS used to measure changes from baseline pre and post 2 weeks physiotherapy session in knee OA patients after mesenchymal stem cell replacement and on 1 month follow up session.
  The Numeric Pain Rating Scale (NPRS) is the simplest and most commonly used numeric scale to rate the pain from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | WOMAC index used to measure changes from baseline pre and post 2 weeks physiotherapy session in knee OA patients after mesenchymal stem cell replacement and on 1 month follow up session.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is widely used to measure symptoms and physical disability, originally developed for people with OA of the hip or knee. It evaluates three dimensions: pain, stiffness, and physical function with 5, 2, and 17 questions. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function, a total of 96, 0 (no symptoms/no limitation) and 96 (maximal symptoms/maximal limitation).
Goniometer (range of motion) | baseline pre and post 2 weeks physiotherapy session in knee OA patients after mesenchymal stem cell replacement and on 1 month follow up session.
  Knee flexion and extension ranges were taken using goniometer to measure changes in ROM.
SF-12 (quality of life) | SF-12 used to measure changes from baseline pre and post 2 weeks physiotherapy session in knee OA patients after mesenchymal stem cell replacement and on 1 month follow up session.
  The SF-12 focuses on patient-based assessments of physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less on the PCS-12 has been recommended as a cut-off to determine a physical condition; while a score of 42 or less on the MCS-12 may be indicative of 'clinical depression.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Institute of Regenerative medicine, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No